CLINICAL TRIAL: NCT04579640
Title: Phase 3 Randomised Controlled Trial of Vitamin D Supplementation to Reduce Risk and Severity of COVID-19 and Other Acute Respiratory Infections in the UK Population
Brief Title: Trial of Vitamin D to Reduce Risk and Severity of COVID-19 and Other Acute Respiratory Infections
Acronym: CORONAVIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other); Pharma Nord (Industry); Fischer Family Trust (Unknown); The AIM Foundation (Unknown); Synergy Biologics Ltd (Unknown); Cytoplan Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 289515
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Acute Respiratory Tract Infection
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Standard of care (national recommendation of 400 IU/day vitamin D)
- Intervention: Lower-dose vitamin D (Experimental): Offer of a daily dose of 800 IU (20 micrograms) cholecalciferol to individuals with 25-hydroxyvitamin D level <75 nmol/L
  Interventions: Dietary Supplement: Vitamin D
- Intervention: Higher-dose vitamin D (Experimental): Offer of a daily dose of 3200 IU (80 micrograms) cholecalciferol to individuals with 25-hydroxyvitamin D level <75 nmol/L
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Capsules containing 800 IU (20 micrograms) or 3,200 IU (80 micrograms) cholecalciferol
  Arms: Intervention: Higher-dose vitamin D; Intervention: Lower-dose vitamin D

SUMMARY:
CORONAVIT is an open-label, phase 3, randomised clinical trial testing whether implementation of a test-and-treat approach to correction of sub-optimal vitamin D status results in reduced risk and/or severity of COVID-19 and other acute respiratory infections.

ELIGIBILITY:
Inclusion criteria:

1. UK resident
2. Age ≥16 years
3. Gives informed consent to participate

Exclusion criteria:

1. taking digoxin, alfacalcidol, calcitriol, dihydrotachysterol or paricalcitol
2. known diagnosis of sarcoidosis, primary hyperparathyroidism, renal stones or renal failure requiring dialysis
3. known allergy to any ingredient in the study capsules (vitamin D, olive oil, caramel, gelatine or glycerol)
4. pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6200 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants experiencing at least one doctor-diagnosed or laboratory-confirmed acute respiratory infection of any cause. | Over 6 months

SECONDARY OUTCOMES:
Proportion of participants developing PCR- or antigen test-positive COVID-19 | Over 6 months
  Secondary efficacy outcome
Proportion of participants who are prescribed one or more courses of antibiotic treatment for acute respiratory infection | Over 6 months
  Secondary efficacy outcome
Proportion of participants with asthma who experience one or more exacerbations of asthma requiring treatment with oral corticosteroids and/or requiring hospital treatment | Over 6 months
  Secondary efficacy outcome
Proportion of participants with COPD who experience one or more exacerbations of COPD requiring treatment with oral corticosteroids and/or antibiotics, and/or requiring hospital treatment | Over 6 months
  Secondary efficacy outcome
Proportion of participants who have had PCR-, antigen test- or antibody test-confirmed SARS-CoV-2 infection who report symptoms of COVID-19 lasting more than 4 weeks after onset | Over 6 months
  Secondary efficacy outcome
Mean MRC dyspnoea score at the end of the study in people who have had PCR-, antigen test- or antibody test-confirmed SARS-CoV-2 infection and who report symptoms of COVID-19 lasting more than 4 weeks after onset | 6 months
  Secondary efficacy outcome
Mean FACIT Fatigue Scale score at the end of the study in people with antigen test- or antibody test-confirmed SARS-CoV-2 infection and who report symptoms of COVID-19 lasting more than 4 weeks after onset | 6 months
  Secondary efficacy outcome
Mean COVID-19 Recovery Questionnaire score at the end of the study in people who have had antigen test- or antibody test-confirmed SARS-CoV-2 infection and who report symptoms of COVID-19 lasting more than 4 weeks after onset | 6 months
  Secondary efficacy outcome
Proportion of participants who experience one or more acute respiratory infections requiring hospitalisation | Over 6 months
  Secondary efficacy outcome
Proportion of participants who experience COVID-19 requiring hospitalisation | Over 6 months
  Secondary efficacy outcome
Proportion of participants hospitalised for COVID-19 requiring ventilatory support | Over 6 months
  Secondary efficacy outcome
Proportion of participants dying of any cause during participation in the trial | Over 6 months
  Secondary efficacy outcome
Proportion of participants dying of acute respiratory infection during participation in the trial | Over 6 months
  Secondary efficacy outcome
Proportion of participants dying of COVID-19 during participation in the trial | Over 6 months
  Secondary efficacy outcome
Mean end-study 25(OH)D concentration (sub-set of participants having end-study tests of vitamin D status) | 6 months
  Secondary efficacy outcome
Proportion of participants experiencing known hypercalcaemia | Over 6 months
  Secondary safety outcome
Proportion of participants experiencing a probable or definite adverse reaction to vitamin D supplementation | Over 6 months
  Secondary safety outcome
Proportion of participants experiencing a serious adverse event of any cause | Over 6 months
  Secondary safety outcome
Proportion of SARS-CoV-2 vaccinated participants with antibodies to SARS-CoV-2 spike protein | Over 6 months
  Secondary efficacy outcome
Median titre of antibodies to SARS-CoV-2 spike protein in SARS-CoV-2 vaccinated participants | Over 6 months
  Secondary efficacy outcome
Proportion of SARS-CoV-2 vaccinated participants with antigen-specific T cell responses to SARS-CoV-2 spike protein (sub-set of participants) | Over 6 months
  Secondary efficacy outcome
Frequency of antigen-specific T cells reacting to SARS-CoV-2 spike protein in SARS-CoV-2 vaccinated participants (sub-set of participants) | Over 6 months
  Secondary efficacy outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, County (optional), United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with other researchers subject to terms of Data Transfer Agreement and IRB approval
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Jolliffe DA, Holt H, Greenig M, Talaei M, Perdek N, Pfeffer P, Vivaldi G, Maltby S, Symons J, Barlow NL, Normandale A, Garcha R, Richter AG, Faustini SE, Orton C, Ford D, Lyons RA, Davies GA, Kee F, Griffiths CJ, Norrie J, Sheikh A, Shaheen SO, Relton C, Martineau AR. Effect of a test-and-treat approach to vitamin D supplementation on risk of all cause acute respiratory tract infection and covid-19: phase 3 randomised controlled trial (CORONAVIT). BMJ. 2022 Sep 7;378:e071230. doi: 10.1136/bmj-2022-071230. PMID 36215226
- See also: Pre-print — https://doi.org/10.1101/2022.03.22.22271707